CLINICAL TRIAL: NCT03831932
Title: A Phase Ib Study of Osimertinib (AZD9291) and Telaglenastat (CB-839) HCl in Patients With EGFR Mutant Non-Small Cell Lung Cancer
Brief Title: Telaglenastat Hydrochloride and Osimertinib in Treating Patients With EGFR-Mutated Stage IV Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00572; NCI-2019-00572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 19016; 10216 (Other: Ohio State University Comprehensive Cancer Center LAO); 10216 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; osimertinib; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (telaglenastat HCl, osimertinib) (Experimental): Patients receive telaglenastat hydrochloride PO BID and osimertinib PO QD (starting cycle 1 day 16 of phase I). Patients undergo blood sample collection and may undergo x-ray imaging, CT scan, MRI, or PET scan throughout the study. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Elastography; Drug: Osimertinib; Procedure: Positron Emission Tomography; Drug: Telaglenastat Hydrochloride; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Telaglenastat Hydrochloride — Given PO
  Other Names: CB-839 HCl; Glutaminase Inhibitor CB-839 Hydrochloride
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase Ib trial studies the side effects and best dose of telaglenastat hydrochloride when given together with osimertinib in treating patients with stage IV non-small cell lung cancer and a mutation in the EGFR gene. Telaglenastat hydrochloride and osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I.To assess the safety and tolerability of osimertinib (AZD9291) and telaglenastat (CB-839) hydrochloride (HCl) and determine the recommended phase II dose (RP2D) in patients with metastatic, EGFR activating mutation-positive non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To determine toxicity profile of the combination of osimertinib (AZD9291) and telaglenastat (CB-839) HCl in patients with metastatic EGFR activating mutation positive NSCLC.

II. To assess the pharmacokinetics (PK) of telaglenastat (CB-839) HCl and osimertinib (AZD9291) in patients with metastatic EGFR activating mutation positive NSCLC.

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. To determine the progression free survival (PFS) of osimertinib (AZD9291) and telaglenastat (CB-839) HCl in patients with EGFR mutation positive NSCLC who have developed progressive disease (PD) on front-line EGFR inhibitor therapy.

II. To determine the overall survival (OS) of osimertinib (AZD9291) and telaglenastat (CB-839) HCl in patients with EGFR mutation positive NSCLC who have developed PD on front-line EGFR inhibitor therapy.

III. To assess cell-free deoxyribonucleic acid (DNA) (cfDNA) and measure changes with response to treatment as well as disease progression (EGFR sensitizing mutations, T790M resistance mutation, recognized bypass mechanisms).

IV. To assess circulating levels of glutamine, glutamate, aspartate and asparagine, and measure changes with response to treatment as well as disease progression.

V. To assess 18F-fluorodeoxyglucose (18F-FDG)-positron emission tomography (PET) parameters at baseline and after treatment to evaluate changes with response to treatment as well as emergence of disease resistance or progression. (Expansion cohort, select patients only)

VI. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing (RNAseq), in order to:

VIa. To identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned.

VIb. To identify resistance mechanisms using genomic DNA- and RNA-based assessment platforms.

OUTLINE: This is a phase I, dose-escalation study of telaglenastat hydrochloride followed by a dose-expansion study.

Patients receive telaglenastat hydrochloride orally (PO) twice daily (BID) and osimertinib PO once daily (QD) (starting cycle 1 day 16 of phase I). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and may undergo x-ray imaging, computed tomography (CT) scan, magnetic resonance imaging (MRI), or positron emission tomography (PET) scan throughout the study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, stage IV NSCLC, with advanced or metastatic disease
* Activating mutation present in the EGFR gene (L858R or exon 19 deletion, alone or in combination with other EGFR mutations) as per local assessment of a tissue biopsy/cytology specimen. The tissue biopsy must have been obtained since the time of disease progression on most recent targeted therapy. "Liquid" biopsies (i.e. blood based) biopsies cannot be used for eligibility determination
* Patients must have had progressive disease on prior EGFR inhibitor therapy (gefitinib, erlotinib, afatinib, or osimertinib). There is no limit to lines of prior tyrosine kinase inhibitor (TKI) therapy. Prior osimertinib (AZD9291) therapy is permitted
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Age > 18 years. NSCLC is exceedingly rare in patients < 18 years of age. Because no dosing or adverse event (AE) data are currently available on the use of telaglenastat (CB-839) HCl in combination with osimertinib (AZD9291) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Must be able to swallow pills
* Life expectancy > 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90 g/L
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) and up to 3 mg/dL for patients with Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN and =< 5 x institutional ULN for patients with liver metastases
* Creatinine within 1.5 x ULN OR
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (measured or calculated by Cockcroft and Gault equation) - confirmation of creatinine clearance is only required for patients with creatinine levels above institutional upper limit of normal
* Should participants with hepatitis B virus (HBV) infection be included, patients are only eligible if they meet all the following criteria:

  * Demonstrated absence of hepatitis C virus (HCV) co-infection or history of HCV co-infection
  * Demonstrated absence of human immunodeficiency virus (HIV) infection
  * Participants with active HBV infection are eligible if they are:

    * Receiving anti-viral treatment for at least 6 weeks prior to study treatment, HBV DNA is suppressed to <100 IU/mL and transaminase levels are below ULN. Participants with a resolved or chronic infection HBV are eligible if they are:

      * Negative for hepatitis B surface antigen (HBsAg) and positive for hepatitis B core antibody [anti-HBc IgG]. In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (To be determined [TBD] by hepatologist) post treatment OR
      * Positive for HBsAg, but for > 6 months have had transaminases levels below ULN and HBV DNA levels below <100 IU/mL (i.e., are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (TBD by hepatologist) post treatment
* If history of hepatitis C virus (HCV) infection, must be treated and have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS) - directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy. Patients on corticosteroids for the treatment of brain metastases will be permitted as long as the dose is =< 10 mg of prednisone-equivalent and has not been increased within 2 weeks of screening
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* EXPANSION COHORT: Patients must have had progressive disease on prior first line EGFR inhibitor therapy with osimertinib

Exclusion Criteria:

* Patients who have not recovered from AEs due to prior systemic anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia. Note: Subjects with irreversible toxicity that in the opinion of the treating physician is not reasonably expected to be exacerbated by the investigational treatment may be included (e.g., hearing loss, hormone deficiency requiring replacement therapy)
* Previous enrollment in the present study
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease
* Patients who are receiving any other investigational agent within five half-lives of the compound or 3 months, whichever is greater. Patients who have received prior immunotherapy may be included only if time from last immunotherapy is at least 3 months (i.e. 90 days)
* Spinal cord compression, symptomatic and unstable brain metastases except for those patients who have completed definitive therapy, and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients may be on corticosteroids (=< 10 mg of prednisone-equivalent) to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic
* Patients with an uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to telaglenastat (CB-839) HCl, osimertinib (AZD9291), or other agents used in study. Patients with hypersensitivity to to any of the inactive excipients thereof should also be excluded
* Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (wash-out periods vary). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
* Pregnant women are excluded from this study because telaglenastat (CB-839) HCl is a glutaminase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with telaglenastat (CB-839) HCl and osimertinib (AZD9291), breastfeeding should be discontinued if the mother is treated with telaglenastat (CB-839) HCl and osimertinib (AZD9291). Breastfeeding patients will be excluded. These potential risks may also apply to other agents used in this study
* Patients with a significant history of cardiovascular disease (e.g., myocardial infarction [MI], thrombotic or thromboembolic event in the last 6 months)
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc using Fridericia's formula [QTcF]) > 470 msec (Fridericia's Criteria for Corrected QT interval [QTc] Calculation: Fridericia's formula QTcF = (QT/RR 0.33). RR is the time from the interval of 1 QRS complex to the next measured in seconds and is commonly calculated as (60/HR)
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < lower limit of normal (LLN); serum/plasma magnesium < LLN; serum/plasma calcium < LLN , congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
  * Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) as assessed by either multigated acquisition (MUGA) scan or echocardiogram (ECHO)
* Patients with active malignancies other than NSCLC or patients with prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers, ductal carcinoma in-situ (DCIS), or indolent cancer currently on observation (i.e. chronic lymphocytic leukemia [CLL] or low-risk prostate cancer)
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection with human immunodeficiency virus (HIV). Screening for chronic conditions is not required
* Patients with symptomatic CNS metastases who are neurologically unstable
* Patients who are at risk for impaired absorption of oral medication including, but not limited to, refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of telaglenastat (CB-839) HCl and osimertinib (AZD9291)
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2026-03-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight H Owen, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant enrolled to be a part of the phase 1b dose escalation but withdrew from the study prior to being assigned to a dose level.
Groups:
- Phase 1b 400mg Telaglenastat HCl Cohort; Phase 1b 600mg Telaglenastat HCl Cohort; Phase 1b 800mg Telaglenastat HCl Cohort; Phase 2 Expansion Cohort: Patients receive telaglenastat hydrochloride PO BID and osimertinib PO QD (starting cycle 1 day 16 of phase I). Patients undergo blood sample collection and may undergo x-ray imaging, CT scan, MRI, or PET scan throughout the study. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT scan
  Magnetic Resonance Elastography: Undergo MRI
  Osimertinib: Given PO
  Positron Emission Tomography: Undergo PET scan
  Telaglenastat Hydrochloride: Given PO
  X-Ray Imaging: Undergo x-ray imaging
Period: Overall Study
Arm/Group | Phase 1b 400mg Telaglenastat HCl Cohort | Phase 1b 600mg Telaglenastat HCl Cohort | Phase 1b 800mg Telaglenastat HCl Cohort | Phase 2 Expansion Cohort
Started | 3 | 3 | 6 | 10
Completed | 3 | 3 | 6 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b 400mg Telaglenastat HCl Cohort | Phase 1b 600mg Telaglenastat HCl Cohort | Phase 1b 800mg Telaglenastat HCl Cohort | Phase 2 Expansion Cohort | Total
Number analyzed (Participants) | 3 | 3 | 6 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 6 | 10
  >=65 years | 2 | 1 | 5 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7 | 14
  Male | 1 | 1 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 5 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 3 | 3
  White | 3 | 3 | 6 | 6 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D)
Time Frame: Up to 28 days
Population: The recommended phase II dose was determined during the phase 1b portion of the study, so only participants from the phase 1b cohorts are included for analysis.
Measure: Number; unit: milligrams
Groups:
- Phase 1b Cohorts: Patients receive telaglenastat hydrochloride PO BID and osimertinib PO QD (starting cycle 1 day 16 of phase I). Patients undergo blood sample collection and may undergo x-ray imaging, CT scan, MRI, or PET scan throughout the study. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Biospecimen Collection: Undergo blood sample collection
  Computed Tomography: Undergo CT scan
  Magnetic Resonance Elastography: Undergo MRI
  Osimertinib: Given PO
  Positron Emission Tomography: Undergo PET scan
  Telaglenastat Hydrochloride: Given PO
  X-Ray Imaging: Undergo x-ray imaging
Arm/Group | Phase 1b Cohorts
Number analyzed (Participants) | 12
milligrams
  Telaglenastat (CB-839) HCl | 800
  Osimertinib (AZD9291) | 80

2. Secondary Outcome: Dose Limiting Toxicities (DLT)
Description: Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: Up to 28 days
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Survival will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Time Frame: From initiation of therapy to documented progression or death without progression, assessed up to 30 days after completion of therapy
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 3
Time Frame: From initiation of therapy to death from any cause, assessed up to 30 days after completion of therapy
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Post-glutaminase Inhibitor CB-839 Hydrochloride Pharmacokinetics (PK) (CB-839 HCl)
Description: Will be assessed by CB-839 HCl drug levels following both single agent therapy as well as combination therapy with CB-839 HCl and osimertinib (AZD9291). Will explore PK endpoints such as concentration steady state (Css), area under the curve (AUC), clearance (CL), volume of distribution (Vd), and half-life (t1/2) computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, generalized estimating equations [GEE]) to assess the PK and pharmacodynamics (PD) markers described above in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.
Time Frame: Day 15 of cycle 1, day 2 of cycle 2 and day 1 of each subsequent cycle (each cycle = 28 days)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Post-AZD9291 Pharmacokinetics
Description: Will be assessed by AZD9291 drug levels following combination therapy with CB-839 HCl and AZD9291. Will be assessed by CB-839 HCl drug levels following both single agent therapy as well as combination therapy with CB-839 HCl and AZD9291. Will explore PK endpoints such as Css, AUC, CL, Vd, and t1/2 computed using non-compartmental and compartmental methods. Will use graphical analyses as well as repeated measure models (linear or nonlinear mixed models, GEE) to assess the PK and PD markers described above in relation to clinical treatment outcomes, recognizing some inherent limitations due to sample size.
Time Frame: Day 2 of cycle 2 and day 1 of each subsequent cycle (each cycle = 28 days)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in EGFR Mutational Status
Description: Will be assessed by cell-free deoxyribonucleic acid (cfDNA). All continuous measurements will be summarized using mean +/- standard error of mean (SEM), range, and median at each time point. Changes in these measurements from baseline to after treatment, or baseline to progression will be assessed using paired Wilcoxon tests. Adjustments for multiple comparisons or multiple outcomes will be performed using Bonferroni correction.
Time Frame: Baseline up to disease progression, assessed up to 30 days after completion of therapy
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Circulating Levels of Glutamine, Glutamate, Aspartate, and Asparagine
Description: Will be assessed by plasma concentrations of these compounds. All continuous measurements will be summarized using mean +/- SEM, range, and median at each time point. Changes in these measurements from baseline to after treatment, or baseline to progression will be assessed using paired Wilcoxon tests. Adjustments for multiple comparisons or multiple outcomes will be performed using Bonferroni correction.
Time Frame: Baseline up to time of disease progression, assessed up to 30 days after completion of therapy
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in 18F-fluorodeoxyglucose (18F-FDG)-Positron Emission Tomography (PET) Imaging
Description: Will be summarized using mean +/- SEM, range, and median. The changes in the FDG-PET/computed tomography (CT) parameter measurements from baseline to after treatment will be compared between responders and non-responders using two sample t-test or Wilcoxon test, whichever is appropriate.
Time Frame: Baseline up to 2 cycles of treatment (each cycle = 28 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Phase 1b 400mg Telaglenastat HCl Cohort | Phase 1b 600mg Telaglenastat HCl Cohort | Phase 1b 800mg Telaglenastat HCl Cohort | Phase 2 Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 0/6 | 2/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/6 | 1/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b 400mg Telaglenastat HCl Cohort (N=3) | Phase 1b 600mg Telaglenastat HCl Cohort (N=3) | Phase 1b 800mg Telaglenastat HCl Cohort (N=6) | Phase 2 Expansion Cohort (N=10)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary duct dilation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-Glutamyl Transferase (GGT) increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b 400mg Telaglenastat HCl Cohort (N=3) | Phase 1b 600mg Telaglenastat HCl Cohort (N=3) | Phase 1b 800mg Telaglenastat HCl Cohort (N=6) | Phase 2 Expansion Cohort (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry heaves (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (1) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing Lights during first dose (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Costolchondritis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gum sensitivity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron deficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sensitive to light (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal flutter (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
altered mental status (intermittent) (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cjills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
creatine phosphokinase (CPK) increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry nares (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontnence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
mouth ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03831932/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03831932/ICF_001.pdf